CLINICAL TRIAL: NCT04373655
Title: A Prospective Multicenter Cohort Study to Evaluate Different Surgical Methods of Axillary Staging (sentinel Lymph Node Biopsy, Targeted Axillary Dissection, Axillary Dissection) in Clinically Node-positive Breast Cancer Patients Treated with Neoadjuvant Chemotherapy
Brief Title: AXillary Surgery After NeoAdjuvant Treatment
Acronym: AXSANA
Status: Recruiting | Type: Observational
Sponsor: European Breast Cancer Research Association of Surgical Trialists (Network)
Collaborators: AWOgyn (Other); AGO-B (Unknown); North Eastern German Society of Gynaecological Oncology (Other); GBG Forschungs GmbH (Other); Claudia von Schilling Foundation for Breast Cancer Research (Unknown); Ehmann-Stiftung Savognin (Unknown)
Responsible Party: Sponsor
Other Study IDs: EUBREAST 3
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant chemotherapy; axillary lymph node dissection; targeted axillary dissection; target lymph node; sentinel node biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The optimal surgical axillary staging technique in patients who convert from the clinically positive to clinically negative lymph node status under neoadjuvant therapy (cN+ → ycN0) remains to be clarified. Different strategies (axillary lymph node dissection, sentinel node biopsy, targeted axillary dissection) are currently used in different countries. A prospective analysis comparing these techniques regarding feasibility, safety, morbidity and surgical effort is urgently needed. Due to high complexity and discordant recommendations, a randomized trial comparing different techniques is hardly feasible. Therefore, the EUBREAST study group decided to initiate a prospective cohort study as an international project that aims at comparatively evaluating data on axillary staging after neoadjuvant therapy.

DETAILED DESCRIPTION:
For many decades, axillary lymph node dissection (ALND) has been considered standard of care in breast cancer (BC) patients. The procedure aimed at assessing the pN status to guide adjuvant therapy decisions as well as ensuring adequate locoregional control. However, ALND is associated with high morbidity and may therefore lead to reduced quality of life in BC patients.

In women undergoing primary surgery, ALND as a staging tool has been replaced by the less invasive sentinel lymph node biopsy (SLNB) without compromising the disease-free or overall survival (DFS, OS). Since then, the therapeutic benefit of ALND in patients with clinically occult metastasis in the sentinel lymph node (SLN) has been challenged as well. According to the current national and international guidelines (e.g. ESMO, NCCN, German S3 guideline and AGO recommendations) completion ALND can be safely omitted in selected patients with 1-2 positive sentinel lymph nodes.

The feasibility and safety of the SLNB after neoadjuvant chemotherapy (NACT) has been controversially discussed, particularly regarding women who initially presented with positive lymph nodes (cN+) and converted to ycN0 following NACT. In these patients, two large prospective multicenter trials reported a false-negative rate (FNR) of 12 and 14%, respectively, thus exceeding the generally accepted (albeit arbitrarily chosen) cutoff of 10%. The clinical relevance of an FNR > 10% and its impact on oncological endpoints (DFS, OS) remains unclear. For this reason, numerous national guidelines still recommend ALND in these patients.

Possible ways to further reduce the FNR in cN+ patients have been extensively discussed in the recent years. In 2016, a novel surgical approach (TAD = targeted axillary dissection) has been reported that consists of inserting a marking (e.g. a clip or a radioactive tracer) into the metastatic lymph node before NACT. In patients in whom the marked lymph node (target lymph node = TLN) and the sentinel node had been successfully removed, the FNR was as low as 1.4%. These retrospectively analyzed data from a prospective register support the hypothesis that TAD can improve the relatively low success rates of SLNB and reduce the long-term morbidity of patients undergoing axillary surgery in the neoadjuvant setting.

Several issues regarding currently used axillary staging techniques remain yet to be clarified. Based on the unclear evidence, the guideline recommendations for the cN+ → ycN0 patients differ strongly. The current ESMO guidelines state that (1) SLNB may be carried out in selected cases, and, if negative, further axillary surgery may be avoided and (2) the FNR of SLNB alone can be improved by marking the biopsied positive node(s) to verify the removal. In Germany, the S3 guideline (last version: 2020) recommends ALND in patients with initial nodal involvement. In contrast, the German Working Group Gynecological Oncology (AGO) changed their recommendations in 2019 and endorsed TAD as a technique of choice for this patient subgroup. In several European countries (Sweden, Norway, Finland) ALND is still considered standard of care for these patients. In others, such as Italy, most patients receive SLNB alone without marking and removing the target lymph node. In the current NCCN guidelines the TAD is considered an optional technique. A prospective analysis comparing different techniques regarding feasibility, safety, morbidity and surgical effort is urgently needed. Due to high complexity and discordant recommendations, a randomized trial comparing different techniques is hardly feasible and therefore would not clarify currently open issues within a reasonable timeframe.

Based on the lack of sufficient evidence and discrepancies between different national and institutional standards, the EUBREAST study group (www.eubreast.com) decided to initiate a prospective cohort study as an international project that aims at comparatively evaluating data on axillary staging after NACT.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Primary invasive breast cancer (confirmed by core biopsy)
* cN+
* cT1-4c
* Scheduled for neoadjuvant systemic therapy
* Female / male patients ≥ 18 years old

Exclusion criteria

* Distant metastasis
* Recurrent breast cancer
* Inflammatory breast cancer
* Extramammary breast cancer
* Supraclavicular lymph node metastasis
* Pregnancy
* Less than 4 cycles of NACT administered
* Patients not suitable for surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with lymph node metastasis undergoing neoadjuvat chemotherapy.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (iDFS) | 5 years
  iDFS is defined as time from surgery to the first clinical, radiological or histological diagnosis of invasive relapse
Axillary recurrence rate | 3 years
  Axillary recurrence is defined as radiological and/or histological diagnosis of tumor recurrence in the axilla
Health-related quality of life | 5 years
  Health-related QoL will be assessed with the EORTC Quality of life questionnaires
Arm morbidity | 5 years
  Arm morbidity will be assessed with the Lymph IFC questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Kühn, Prof., Study Chair — European Breast Cancer Research Association of Surgical Trialists
Locations (1):
- Klinikum Esslingen, Esslingen am Neckar, Germany

REFERENCES:
- [Derived] Banys-Paluchowski M, Hartmann S, Basali T, Gasparri ML, de Boniface J, Gentilini OD, Cakmak GK, Ditsch N, Stickeler E, Schlichting E, Rubio I, Peintinger F, Untch M, Mau C, Federspiel FK, Bucher S, Ramaker K, Paluchowski P, Bauer L, Riemer S, Langanke D, Leuf TD, Schnabel J, von Abel E, Solbach C, Ovalle SC, Hilmer K, Bjelic-Radisic V, Stahl N, Sanchez-Mendez JI, Hagen V, Hansen MH, Krawczyk N, Sezen BA, Jursik K, Thill M, Kolberg HC, Reimer T, Ruf F, Wihlfahrt K, Rief A, Berger T, Schmidt E, Tauber N, Frohlich S, Kuhn T. Radar reflectors for marking of target lymph nodes in initially node-positive patients receiving neoadjuvant chemotherapy for breast cancer-a subgroup analysis of the prospective AXSANA (EUBREAST-03) trial. Breast Cancer Res Treat. 2025 May;211(1):203-211. doi: 10.1007/s10549-025-07635-4. Epub 2025 Feb 20. PMID 39976867
- [Derived] Hartmann S, Banys-Paluchowski M, Stickeler E, de Boniface J, Gentilini OD, Kontos M, Seitz S, Kaltenecker G, Warnberg F, Zetterlund LH, Kolberg HC, Frohlich S, Kuhn T. Applicability of magnetic seeds for target lymph node biopsy after neoadjuvant chemotherapy in initially node-positive breast cancer patients: data from the AXSANA study. Breast Cancer Res Treat. 2023 Dec;202(3):497-504. doi: 10.1007/s10549-023-07100-0. Epub 2023 Sep 8. PMID 37684426